CLINICAL TRIAL: NCT02309814
Title: Eyelid Movement Sensor Device- Blinking Characterizing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, daniel briscoe, Head of ophthalmology departement, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0133-13-EMC
Record Dates: First submitted 2014-12-01; First posted 2014-12-05 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Eyelid Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eyelid motion sensor device (Experimental): all volunteers will wear the monitor eyelid sensor device (including the tiny magnets on the upper eyelid). a 10 minutes movie will be screened on 40 inch television screen in a 3 meters distance.
  Interventions: Device: eyelid motion sensor device (Hall-probe)

INTERVENTIONS:
Device: eyelid motion sensor device (Hall-probe) — all volunteers will wear the eyelid motion sensor device (Hall-probe) (including the tiny magnets on the upper eyelid). a 10 minutes movie will be screened on 40 inch television screen in a 3 meters distance

SUMMARY:
The investigators have developed a simple to use device that facilitates the monitoring of the upper eyelids motion, acquires the eyelid vertical movement and enables analysis and graphic presentation of the results. the device system consists 3 components : glasses for the patient including magneto sensitive probes, hardware and dedicated software.

Our purpose is to characterize eyelid motion in normal population. The methods include measuring each patient 10 minutes during watching a short movie.

DETAILED DESCRIPTION:
Essentially, for Hall-probes monitor the magnetic field generated by a tiny magnets attached to the upper eyelid.

ELIGIBILITY:
Inclusion Criteria:

* healthy 18-67 year olds with no eye medical history

Exclusion Criteria:

* pregnancy
* head trauma history
* using contact lens

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Demonstrate and describe measurable blinking character in normal population.(Hall-probes monitor the magnetic field generated by a tiny magnets attached to the upper eyelid) | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: daniel briscoe, Principal Investigator — haemek medical center